CLINICAL TRIAL: NCT00481468
Title: Validation of the Siemens System Somatom Definition and Operating Software SYNGO CT2007 (Software Version SOMARIS/7 SYNGO® Software) for Cardiac CT Studies
Brief Title: Validation of the Siemens System Somatom Definition and Operating Software for Cardiac CT Studies
Acronym: SOMARIS
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Gilbert L. Raff, MD, Medical Director of Advanced Cardiovascular Imaging, Corewell Health East
Other Study IDs: 2006-059
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Chest Pain
Keywords: Coronary artery disease; chest pain
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We are evaluating a new computer software package to help us acquire and interpret heart CT studies, which is the purpose of this research project. We plan to compare the acquiring and analysis of heart artery calcium scores and CT angiograms (scans of the heart arteries) with the new SYNGO Somaris/7 Cardiac software to our previous experience with the the existing Siemens software and the TeraRecon software (current software used in the Cardiovascular MR/CT lab). The main objective of this study is to provide information to Siemens regarding the ease of use and capability of the scanner's software. The goal of this study is to determine whether the acquisition and interpretation information with the new software functionally meets the guidelines specified by Siemens, and also to determine whether the software is equivalent or superior to previous versions we used from April 2004 to April 2006.

DETAILED DESCRIPTION:
We will obtain and read CT coronary angiograms (CAT scans of the heart arteries) with the assistance of the new imaging software analysis package. Analysis of technical and clinical data will be recorded on the case report forms. This will be an observational design. We intend to test the results of our analyses through a Test Plan looking at Cardio functionality (hardware and software), System performance (reconstruction, loading, transferring, archiving),and System stability.

We plan to find out the relevant effect of our clinical reading results by enrolling our patients in a long-term clinical outcomes database. To evaluate the presence of traditional coronary risk factors, a focused medical history will be requested (see attached) as well as access to relevant medical records to determine the presence of major adverse cardiac events. These will be handled in a confidential manner and will be de-identified using subject number and initial only to be compliant with HIPAA.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. Age equal to or greater than 18 years -

Exclusion Criteria:

1. Renal (kidney) insufficiency (creatinine greater than or equal to 1.6) or renal (kidney) failure requiring dialysis.
2. Atrial fibrillation (type of heart rhythm) or other markedly irregular rhythm.
3. Inability or refusal to provide informed consent.
4. Psychological unsuitability or extreme claustrophobia (fear of closed in spaces).
5. Pregnancy or unknown pregnancy status.
6. Age less than 18 years.
7. Clinical instability as deemed by the attending physician, including cardiogenic shock, hypotension (low blood pressure-systolic blood pressure less than 90 mmHg), refractory hypertension (high blood pressure) (systolic blood pressure greater than 180 mmHg), sustained ventricular or atrial arrhythmia (types of heart rhythm) requiring intravenous medications.
8. Inability to tolerate beta-blockers, including those with chronic obstructive pulmonary disease (temporary narrowing of the tubes in the lungs) (or asthma requiring maintenance inhaled bronchodilators or steroids, complete heart block (chambers in the heart not beating in sync), second-degree atrioventricular block (chambers in the heart not beating in sync).
9. Known contrast dye allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This sutdy is taking place in a 900+ bed community setting hospital. All patients who meet the inclusion and exclusion criteria will be asked if they would like to participate when they arrive to the radiology department to undergo their cornary CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Raff, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States